CLINICAL TRIAL: NCT02277145
Title: Phase I Study of Radiation-induced Pulmonary Fibrosis Treated With Clinical Grade Umbilical Cord Mesenchymal Stem Cells
Brief Title: A Study on Radiation-induced Pulmonary Fibrosis Treated With Clinical Grade Umbilical Cord Mesenchymal Stem Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jianwu Dai (Other Government)
Collaborators: Southwest Hospital, China (Other)
Responsible Party: Sponsor-Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Organization: Chinese Academy of Sciences (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAS-XDA001-SH/IGDB
Record Dates: First submitted 2014-10-20; First posted 2014-10-28 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2018-07

CONDITIONS: Post-radiotherapy Pulmonary Fibrosis
Keywords: radiation-induced pulmonary fibrosis; MSCs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment group (Experimental): Patients will receive 10^6 (1 million) /Kg/person cells of clinical grade umbilical cord mesenchymal stem cells (MSCs) injected via fiberoptic bronchoscopy after fully lavage of the localized lesions
  Interventions: Biological: clinical grade umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: clinical grade umbilical cord mesenchymal stem cells — 10^6 (1 million) /Kg/person cells of clinical grade umbilical cord MSCs will be injected after fully lavage of the localized lesions

SUMMARY:
Radiation therapy is one of the main means for treating malignant tumor, during which radioactive lung injury is inevitable. Currently there is nearly no effective clinical treatment for late post-radiotherapy pulmonary fibrosis. This study intends to carry out an open, single-center, non-randomized phase I clinical trial. During the treatment, the local lesions will be fully lavaged, and then clinical grade umbilical cord mesenchymal stem cells (MSCs) will be injected directly into the lesion by fiberoptic bronchoscopy. After six-month observation, the investigators will initially evaluate the safety and effectiveness of the treatment by measuring two key indicators-the CT density histogram and the patients' self-evaluation, and one secondary indicator-the changes of TGF-β1 contents, both before and after the treatment. Meanwhile, the investigators will make a preliminary discuss about the possible immunomodulatory effects of the umbilical cord MSCs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-70 years old.
2. Subjects with a clear history of malignancy.
3. Subjects with a clear history of chest radiation therapy at least 3 months earlier.
4. Subjects diagnosed as chronic phase of radiation-induced pneumonitis or radiation-induced pulmonary fibrosis stage (see Annex 3 for diagnosis).
5. Subjects signed informed consent.

Exclusion Criteria:

1. Women of childbearing age at the stage of pregnancy or lactation, or those without taking effective contraceptive measures.
2. Subjects with syphilis or HIV positive antibody.
3. Subjects with infection aggravated within the past month.
4. Subjects suffering from any of the following pulmonary diseases: active tuberculosis, pulmonary embolism, pneumothorax, multiple huge bullae, uncontrolled asthma, severe pneumonia, acute exacerbation of chronic bronchitis, AECOPD, severe and / or extremely severe COPD, etc..
5. Subjects suffering from other serious diseases, such as myocardial infarction, unstable angina, cirrhosis, and acute glomerulonephritis.
6. Subjects with progression-free survival (PFS) less than 0.5 years or Karnofsky performance scores less than 60 points.
7. Subjects with leukopenia (WBC less than 4x109 / L) or agranulocytosis (WBC less than 1.5x109 / L or neutrophils less than 0.5x109 / L) caused by any reason.
8. Subjects with severe renal impairment, serum creatinine> 1.5 times the upper limit of normal.
9. Subjects with liver disease or liver damage: ALT, AST, total bilirubin> 2 times the upper limit of normal
10. Subjects with a history of mental illness or suicide risk, with a history of epilepsy or other central nervous system disorders.
11. Subjects with severe arrhythmias (such as ventricular tachycardia, frequent superventricular tachycardia, atrial fibrillation, and atrial flutter, etc.) or cardiac degree II or above conduction abnormalities displayed via 12-lead ECG.
12. Subjects with a history of alcohol or illicit drug abuse.
13. Subjects accepted by any other clinical trials within 3 months before the enrollment
14. Subjects with poor compliance, difficult to complete the study.
15. Any other conditions that might increase the risk of subjects or interfere with the clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Composite indicators, including quantitative analysis of CT density histograms, self-evaluation and changes of TGF-β1 content | 6 months
  Different proportions will be assigned to the three indicators. The overall curative effect can be judged with scores ranging from 0 to100. Specific proportions are as follows: full scores of 50 points for image changes, 25 for self-efficacy evaluation and 25 for TGF-β1 content changes. The image changes can be classified into four levels: significant control, improved, stable, and progressive; the self-efficacy evaluation can also be classified into four levels: effective, improved, stable and invalid; the changes of TGF-β1 content will be classified into three levels: improved, stable, and progressive. The four levels will be scored on the ratio of 5:4:3:1, the three levels will be scored on the ratio of 5:3:1.
Safety Evaluation | 6 months
  Clinical adverse events evaluated as definitely/ probably/possibly concerned with stem cell therapy in this trial and abnormal results of laboratory tests or other special examinations will be observed and recorded in detail.

SECONDARY OUTCOMES:
Clinical Indicator 1: change in blood gas analysis | 3-6 months
Clinical Indicator 2: change in pulmonary function analysis | 3-6 months
Clinical Indicator 3: 6-minute walk test distance | 3-6 months
Clinical Indicator 4: change in MRC chronic dyspnea scale | 3-6 months
Clinical Indicator 5: change in St. George's Respiratory Questionnaire (SGRQ) scale | 3-6 months
Immunological Indicator in serum 1: T lymphocyte counts in peripheral blood | 3-6 months
  Cellular immunological indicator: T lymphocyte counts in peripheral blood measured in serum
Immunological Indicator in serum 2: response level of CD4+ T lymphocyte subsets (such as Th1 / Th2) | 3-6 months
  Cellular immunological indicator: response level of CD4+ T lymphocyte subsets (such as Th1 / Th2) measured in serum
Immunological Indicator in serum 3: concent of immunoglobulin | 3-6 months
  Humoral immunological indicator: concent of immunoglobulin measured in serum
Immunological Indicator in serum 4: expression levels of various cytokines (IL-1, IL-3, IL-6, IL-8, TNF-α, GM-CSF, etc) | 3-6 months
  Humoral immunological indicator: expression levels of various cytokines in serum (IL-1, IL-3, IL-6, IL-8, TNF-α, GM-CSF, etc) measured in serum
Immunological Indicator in serum 5: subtype analysis and phagocytic activity analysis of macrophage | 3-6 months
  Macrophage-related polarization indicator: subtype analysis and phagocytic activity of macrophage measured in serum
Immunological Indicator in serum 6: expression levels of IL-12, IL-10 | 3-6 months
  Macrophage- related polarization indicators: expression levels of IL-12, IL-10 measured in serum
Immunological Indicator in lavage fluid 1: T lymphocyte counts in peripheral blood | 6 months
  Cellular immunological indicator: T lymphocyte counts in peripheral blood measured in lavage fluid
Immunological Indicator in lavage fluid 2: response level of CD4+ T lymphocyte subsets (such as Th1 / Th2) | 6 months
  Cellular immunological indicator: response level of CD4+ T lymphocyte subsets (such as Th1 / Th2) measured in lavage fluid
Immunological Indicator in lavage fluid 3: concent of immunoglobulin | 6 months
  Humoral immunological indicator: concent of immunoglobulin measured in lavage fluid
Immunological Indicator in lavage fluid 4: expression levels of various cytokines (IL-1, IL-3, IL-6, IL-8, TNF-α, GM-CSF, etc) | 6 months
  Humoral immunological indicator: expression levels of various cytokines (IL-1, IL-3, IL-6, IL-8, TNF-α, GM-CSF, etc) measured in lavage fluid
Immunological Indicator in lavage fluid 5: subtype analysis and phagocytic activity analysis of macrophage | 6 months
  Macrophage-related polarization indicator: subtype analysis and phagocytic activity of macrophage measured in lavage fluid
Immunological Indicator in lavage fluid 6: expression levels of IL-12, IL-10 | 6 months
  Macrophage-related polarization indicators: expression levels of IL-12, IL-10 measured in lavage fluid
Inflammatory Indicators: measured by routine blood test including C-reactive protein (CRP) | 3 months
Fibrosis Indicators in serum 1: content of transforming growth factor -α/β (TGF-α/TGF-β) | 3-6 months
  Content of transforming growth factor α/β (TGF-α/TGF-β) measured in serum
Fibrosis Indicators in serum 2: content of hydroxyproline | 3-6 months
  Content of hydroxyproline measured in serum
Fibrosis Indicators in serum 3: content of matrix metalloproteinase 1/7(MMP1/MMP7) | 3-6 months
  Content of matrix metalloproteinase 1/7(MMP1/MMP7) measured in serum
Fibrosis Indicators in lavage fluid 1: content of transforming growth factor -α/β (TGF-α/TGF-β) | 6 months
  Content of transforming growth factor -α/β (TGF-α/TGF-β) measured in lavage fluid
Fibrosis Indicators in lavage fluid 2: content of hydroxyproline | 6 months
  Content of hydroxyproline measured in lavage fluid measured in lavage fluid
Fibrosis Indicators in lavage fluid 3: content of matrix metalloproteinase 1/7(MMP1/MMP7) | 6 months
  Content of matrix metalloproteinase 1/7(MMP1/MMP7) measured in lavage fluid

CONTACTS AND LOCATIONS:
Overall Officials: JianWu Dai, Ph.D, Principal Investigator — Chinese Academy of Sciences; Wei Xiong, M.D, Study Chair — First Affiliated Hospital of the Third Military University, PLA (Southwest Hospital); Xiaotian Dai, M.M, Study Director — First Affiliated Hospital of the Third Military University, PLA (Southwest Hospital)
Locations (1):
- First Affiliated Hospital of the Third Military University, PLA (Southwest Hospital), Chongqing, Chongqing Municipality, China